CLINICAL TRIAL: NCT00197964
Title: A Randomized Trial to Improve Quality of Life Outcomes in Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NHLBI K23 HL 04067
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Asthma
Keywords: Self-management; Self-efficacy; Quality of life; Resource utilization
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Enhance asthma knowledge, self-efficacy, social support

SUMMARY:
Among 180 patients with moderate asthma, the specific aim of this randomized trial is to assess the effectiveness of an intervention involving education, enhancement of self-efficacy, and asthma social support in preventing deterioration in functional status over two years.

DETAILED DESCRIPTION:
The goals of this study are to develop and implement a multi-component intervention to improve quality of life and decrease urgent resource utilization in adult asthma patients followed in a primary care practice. Specifically, the intervention involves a two-component self-directed self-management workbook. The first component focuses on increasing knowledge by providing patients with factual information about asthma and self-management. The second component focuses on asthma self-efficacy using case vignettes and making a contract to adopt a behavior to improve asthma. Asthma-related social support is achieved through interval telephone contact.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for this study if they are 18 years of age or older and have moderate asthma based on the NHLBI Asthma Expert Panel's classification which rates symptoms, frequency of exacerbations, nocturnal attacks, activity restriction, use of medications, and pulmonary function.

Exclusion Criteria:

* Patients will be excluded from this study for the following reasons: if they are have other pulmonary diseases; if they are unable to provide informed consent because of cognitive deficits; if they are not fluent in English; if they refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2001-08; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in the Asthma Quality of Life Questionnaire scores from enrollment to two years.

SECONDARY OUTCOMES:
The secondary outcomes are change in Asthma Self-efficacy Scale scores and differences in urgent resource utilization between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- New York Presbyterian Hospital - Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Background] Mancuso CA, Rincon M, McCulloch CE, Charlson ME. Self-efficacy, depressive symptoms, and patients' expectations predict outcomes in asthma. Med Care. 2001 Dec;39(12):1326-38. doi: 10.1097/00005650-200112000-00008. PMID 11717574
- [Background] Mancuso CA, Peterson MG, Charlson ME. Effects of depressive symptoms on health-related quality of life in asthma patients. J Gen Intern Med. 2000 May;15(5):301-10. doi: 10.1046/j.1525-1497.2000.07006.x. PMID 10840265
- [Background] Mancuso CA, Peterson MG. Different methods to assess quality of life from multiple follow-ups in a longitudinal asthma study. J Clin Epidemiol. 2004 Jan;57(1):45-54. doi: 10.1016/S0895-4356(03)00248-8. PMID 15019010
- [Background] Mancuso CA, Rincon M, Robbins L, Charlson ME. Patients' expectations of asthma treatment. J Asthma. 2003 Dec;40(8):873-81. doi: 10.1081/jas-120023578. PMID 14736086
- [Background] Mancuso CA, Rincon M, Charlson ME. Adverse work outcomes and events attributed to asthma. Am J Ind Med. 2003 Sep;44(3):236-45. doi: 10.1002/ajim.10257. PMID 12929143
- [Result] Mancuso CA, Sayles W, Allegrante JP. Randomized trial of self-management education in asthmatic patients and effects of depressive symptoms. Ann Allergy Asthma Immunol. 2010 Jul;105(1):12-9. doi: 10.1016/j.anai.2010.04.009. PMID 20642198
- [Result] Mancuso CA, Sayles W, Allegrante JP. Knowledge, attitude, and self-efficacy in asthma self-management and quality of life. J Asthma. 2010 Oct;47(8):883-8. doi: 10.3109/02770903.2010.492540. PMID 20831465
- [Derived] Mancuso CA, Sayles W, Allegrante JP. Development and testing of the Asthma Self-Management Questionnaire. Ann Allergy Asthma Immunol. 2009 Apr;102(4):294-302. doi: 10.1016/S1081-1206(10)60334-1. PMID 19441600
- [Derived] Choi TN, Westermann H, Sayles W, Mancuso CA, Charlson ME. Beliefs about asthma medications: patients perceive both benefits and drawbacks. J Asthma. 2008 Jun;45(5):409-14. doi: 10.1080/02770900801971834. PMID 18569235